CLINICAL TRIAL: NCT04321668
Title: A Proof of Concept Study in Patients Suffering of Knee Osteoarthritis (OA) and Receiving Intra-articular (IA) Injection of Synvisc-one® to Assess the Clinical Pertinence of a New Analytical Tool of Synovial Fluid
Brief Title: Innovative Tool to Analyse Synovial Fluid of Patients With Knee Ostearthritis After IA Injection of Synvisc-one®
Acronym: RESYF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulsalys (Industry)
Collaborators: Artialis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RESYF
Record Dates: First submitted 2020-03-10; First posted 2020-03-25 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Knee Osteoarthritis; Intra-Articular Injection
Keywords: Osteoarthritis; food supplement; SYNVISC; Synovial Fluid analysis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Proof of Concept (PoC), monocentric, non-comparative, interventional trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injection of SYNVISC-ONE (Other): Patients suffering from symptomatic knee osteoarthritis (OA), receiving intra-articular (IA) injection of SYNVISC-ONE® (Hylan G-F 20; 10 mL single-injection viscosupplement)
  Interventions: Device: Synvisc-One

INTERVENTIONS:
Device: Synvisc-One — SYNVISC-ONE® (Hylan G-F 20), 10 mL single-injection viscosupplement Status : CE marked (CE 0086) class III Medical Device The IP is used according to its usual dosage, administration and indication
  Other Names: SYNVISC; Hylan G-F 20

SUMMARY:
The objective of this trial is to assess the clinical pertinence of an innovative analytical tool (SYNODIAG) to analyze the Synovial Fluid (SF) composition and guide the patient treatment in a Proof of Concept (PoC) study using OA patients receiving IA injection of SYNVISC ONE®.

DETAILED DESCRIPTION:
In a recent study on animal model (results not yet published), the use of drop deposition combined to Raman spectroscopy provided for the first time the Raman spectral signature of healthy SF. Tribological analysis of simple dried drops of SF showed the potentiality to observe physical and chemical changes due to OA process. HA concentration was correlated with the dried drop area and the increase of protein content was correlated with the height of the peripheral rim. Spectral acquisitions detailed/specified these observations as degradation of cartilage and bone tissues was measured using specific Raman band ratios. These results suggested that DDRS could be an innovative tool in OA clinical research. In this context, the Sponsor would like to assess the clinical pertinence of this innovative analytical tool in a PoC study using OA patients receiving IA injection of SYNVISC ONE®.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 40 years of age with BMI ≤ 35 kg/m2
* Femorotibial knee OA (Uni- or bilateral):

  * Responding to clinical and radiological criteria of American College of Rheumatology (ACR)
  * Symptomatic for more than 6 months in the most painful knee
* Moderate-to-severe knee pain: knee pain score evaluated on VAS (0-100) ≥ 40 over the last month at the inclusion visit (the most painful knee is considered)
* Eligible for knee viscosupplementation using SYNVISC-ONE®
* Knee swelling justifying SF aspiration at baseline - Able to follow the instructions of the study
* Having signed an informed consent

Exclusion Criteria:

1. Related to the OA pathology

   * Recent macro-trauma (< 6 months) of the knee responsible of the symptomatic knee. Micro-trauma are allowed according the Investigator's discretion
   * Concurrent articular disease interfering with the evaluation of OA and/or pain such as but not limited to articular dysplasia, aseptic osteonecrosis, acromegaly, Paget's disease, hemophilia, hemochromatosis, chondromatosis, villonodular synovitis of the knee, seronegative spondyloarthropathy, rheumatoid arthritis, gouty arthritis, infectious arthritis, radiculalgia in the lower limbs, arteritis, chondrocalcinosis x-rays diagnosed and Calcium PyroPhosphate Dihydrate crystal deposition disease (CPPD)
   * Hemarthrosis
   * Prosthesis in the target knee
2. Related to treatment

   * Corticosteroids injection in the target knee in the last 3 months before injection (excepted for low dose injection following SF aspiration at V1 as recommended by standard treatment guidelines)
   * Hyaluronan injection in the target knee in the last 6 months before injection
   * Arthroscopy in the last 3 months before injection
   * Oral corticotherapy ≥ 5mg/day (in Prednisolone equivalent) in the last 3 months before injection
   * Change in the dosage regimen of symptomatic slow-acting drugs for osteoarthritis (SYSADOA) or dietary supplement, i.e., curcuma extract, chondroitin, glucosamine, diacerein or avocado-soya unsaponifiables in the last 3 months before injection
   * An anticipated need for any forbidden OA treatments during the trial
   * Contraindications to SYNVISC-ONE®: hypersensitivity or allergy to the product components and infections or skin diseases in the area of the injection site
   * Anticoagulant anti-vitamin K (such as coumarinic) before injection
3. Related to associated diseases

   * Severe and uncontrolled diseases (type I diabetes, liver failure, renal failure, lung/heart disease, progressive malignant neoplasia or in remission for less than 5 years, HIV)
   * Malignancy or history of malignancy, or other major disease (e.g., systemic fungal infection) or other severe uncontrolled conditions (e.g., drug or alcohol abuse), that are significant and/or that may pose a health risk to the subject in the study or may have an impact on the study assessments
   * High risk of hemorrhage and risk of infection at the site of injection
   * Anticipated need for any surgical or other invasive procedure during the trial including prosthesis in the target knee
4. Related to patients

   * Close collaborators to the Sponsor, the study coordinator or the Investigator
   * Participation in a clinical trial in the last 3 months before injection
   * Patient under guardianship or judicial protection
   * Pregnancy, breastfeeding, planned conception, or premenopausal women without effective contraception (pill, patch, ring, diaphragm, implant and intrauterine device), tubal ligation or hysterectomy
5. Related to MRI counter-indication

   * Risk groups for MRI scanning due to magnetic field: metal in body: pacemaker/AICD/ICD (coronary defibrillator), nervus vagus stimulator, artificial heart valve (depending on type), metal clips on cerebral arteries or veins, metal particles in eye, port-a-cath, metal stents, hydrocephalic pump/insuline pump, metal implants; f/e screws, prostheses, piercings
   * Claustrophobia or serious mobility problem (uncontrolled Parkinson, tremors)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Detection of variation of the composition of Synovial Fluid after hyaluronic acid viscosupplementation in Osteoarthritis patients receiving SYNVISC-ONE® injection | 6 months (between T0 and T6 visit)
  Tribological properties (i.e. the dried drop surface and the peripheral height profile) of the synovial fluid will be analyzed through optical microscopy (2D morphological examinations) in OA patients receiving SYNVISC-ONE® injection

SECONDARY OUTCOMES:
Detection of Synovial fluid tribological properties through interferometry | 6 months (between T0 and T6 visit)
  Topography measurement (3D tribological examination) will be performed using white light interferometry (smartWLI-microscope, GBS mbH, Germany) on the periphery of the drops.
Detection of Synovial fluid molecular structural and chemical changes using a Raman confocal microscope | 6 months (between T0 and T6 visit)
  Based on Raman spectroscopy
Detection of dried drops physicochemical index | 6 months (between T0 and T6 visit)
  Based on surface of dried drops and Raman ratios
Variation of Visual Analogue Scale for the mean knee pain at rest and while walking over the last month | 6 months (between T0 and T6 visit)
  The pain Visual Analogue scale (VAS) is a continuous scale comprised of a horizontal line, usually 10 centimeters in length, anchored by 2 verbal descriptors, one for each symptom extreme.
Variation of Knee injury and Osteoarthritis Outcome Score using a self-administered questionnaire | 6 months (between T0 and T6 visit)
  The KOOS outcome score is a 42-item self-administrated questionnaire comprising 5 subscales: Pain, Symptoms, Activities of Daily Living, Sports and Recreation function, and Quality Of Life. A separate score ranging from 0 to 100, where 100 represents the best result, will be calculated for each subscale. A global score will be calculated by summing the score of each subscale.
Variation of Visual Analogue Scale for patient global assessment of disease activity | 6 months (between T0 and T6 visit)
  The Visual Analogue Scale (VAS) is a continuous scale comprised of a horizontal line, usually 10 centimeters in length, anchored by one verbal descriptors for Global Assessment of disease activity.
Determination of Semi-quantitative Whole ORgan Magnetic Imaging Score score of the joint | At baseline visit (T0)
  MRI Imaging will be analyzed for WORMS by central reading in order to find correlation between the Imaging and the synovial fluid composition.
Responder rate to treatment defined as changes in knee pain and/or knee function and/or patients disease activity according to OMERACT OARSI criteria | 6 months (between T0 and T6 visit)
  Responder criteria for osteoarthritis clinical trials will be based on the questionnaires describe above.
Tolerance to the product | 6 months (between T0 and T6 visit)
  Number of Adverse events (AE or Adverse Device Effect or Device Deficiency; will be coded in terms of SOC and LLT using the last version of MedDRA) and drop offs

OTHER OUTCOMES:
Correlation at each timepoint between Synovial fluid composition and osteoarthritis biological markers (optional) | 6 months (between T0 and T6 visit)
  Monitor the cartilage degeneration by determining the serum level of OA biomarkers through immunoassay (optional)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Emile Dubuc, MD, Principal Investigator — Cliniques Universitaires Saint-Luc UCL
Locations (3):
- Belgium (3):
  - Centre Medical Chant d'Oiseau, Woluwe-Saint-Pierre - Sint-Pieters-Woluwe, Brussels Capital
  - Hopital Delta, CHIREC, Auderghem
  - Cliniques Universitaires Saint Luc - UCL, Woluwe-Saint-Pierre - Sint-Pieters-Woluwe

IPD SHARING:
Plan to Share IPD: No